CLINICAL TRIAL: NCT02233998
Title: 21 Day Clinical Efficacy of Essential Oil Containing Mouth Rinses: Effect on Reducing Existing Gingivitis and Plaque
Brief Title: A Clinical Trial to Test the Effect of Marketed Mouth Rinses on Decreasing Plaque and Gum Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CO-140508133810-OCCT
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Plaque; Gingivitis
Keywords: Plaque; Bleeding; Gums; Gingiva; Gingival Inflammation; Gingival Bleeding
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis; Hemorrhage; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mouth Rinse 1 (Active Comparator): After brushing in your normal manner, rinse full strength twice a day with 20 mL for 30 seconds.
  Interventions: Other: Mouth Rinse 1
- Mouth Rinse 2 (Active Comparator): After brushing in your normal manner, rinse full strength twice a day with 20 mL for 30 seconds.
  Interventions: Other: Mouth Rinse 2
- Mouth Rinse 3 (Placebo Comparator): After brushing in your normal manner, rinse full strength twice a day with 20 mL for 30 seconds.
  Interventions: Other: Mouth Rinse 3

INTERVENTIONS:
Other: Mouth Rinse 1
  Other Names: Cool Mint Listerine Antiseptic
  Arms: Mouth Rinse 1
Other: Mouth Rinse 2
  Other Names: Listerine Zero
  Arms: Mouth Rinse 2
Other: Mouth Rinse 3
  Other Names: Placebo
  Arms: Mouth Rinse 3

SUMMARY:
The reduction of existing plaque and gum inflammation will be evaluated using two marketed mouth rinses along with tooth brushing after 21 days of use compared to a placebo mouth rinse.

165 healthy volunteers will be enrolled in this three week study. Volunteers who qualify to be in this study will have an equal chance of being assigned to one of the three treatment groups. Volunteers will have a total of three visits including 1) Screening/Baseline Day 1 2) Day 11 (after 10 days of use) and 3) Day 22 (after 21 days of use). Volunteers will maintain a diary at home to record each treatment use and will be asked to come to the clinic without brushing or use their product for at least 8 hours, but no more than 18 hours. Examinations for oral hard/soft tissue, gingivitis, bleeding and plaque assessments will be completed at Screening/Baseline and repeated at Clinic Visit 3, which is Day 22.

DETAILED DESCRIPTION:
A sufficient number of generally healthy subjects (approximately 165) that meet the required inclusion/exclusion criteria will be enrolled in this 21 day, examiner-blind, single center, randomized, parallel-group controlled clinical trial to ensure that at least 150 subjects (50 per treatment group) complete this study.

At baseline, the prescreened subjects will present to the clinic site for baseline examinations (oral tissue assessment, gingivitis, bleeding and plaque assessments) having refrained from oral hygiene for at least 8 hours, but no more than 18 hours. After the baseline oral examinations, assessment of other inclusion/exclusion criteria qualifying subjects will be randomly assigned to one of three treatment groups. Immediately following this randomization, subjects will begin use of their assigned test product following the label instructions. If randomized to the control group, subjects will brush twice daily in their usual manner with an ADA accepted fluoride toothpaste and a soft bristled toothbrush followed by rinsing twice daily with a 5% hydroalcohol control rinse (W002194-221P). If randomized to an active treatment group; subjects will brush twice daily in their usual manner, followed by rinsing twice daily with their assigned mouth rinse formulation (19292-116A or 11965-059). Subjects will be instructed to follow label instructions 20ml for 30 seconds twice daily for mouth rinse product. The first product use will be conducted under the supervision of study personnel. All other brushing and rinsing will be unsupervised and the subjects will be required to maintain a diary card to document twice daily product use, brushing and rinsing times. Compliance will be evaluated by weighing residual volumes of returned mouth rinse and by reviewing the subject diary. Subjects will receive an ADA- accepted fluoride-containing dentifrice and a soft bristled toothbrush at their baseline visit.

Subjects may continue to use floss to remove impacted food between the teeth if it is part of their usual oral care regimen during the course of the study; no other oral hygiene procedures will be permitted, including teeth cleaning, whitening or dental procedures except for an emergency treatment. The decision to withdraw a subject due to emergency dental treatment will occur at the discretion of the Investigator.

At baseline and three weeks (±2 days) visits, subject will not have brushed or have used their product for at least 8 hours, but no more than 18 hours.

Oral tissue safety, Modified Gingival Index (MGI), Bleeding Index (BI), and Plaque Index (PI) will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment;
2. Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial;
3. Males and females 18 years of age or older, in good general and oral health without any known allergy to commercial dental products;
4. A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count;
5. A mean gingival index ≥ 1.95 according to the Modified Gingival Index;
6. A mean plaque index ≥ 1.95 according to the Turesky modification of the Quigley-Hein Plaque Index scored on six surfaces per tooth;
7. Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator;
8. Absence of moderate/advanced periodontitis based on a clinical examination (ADA Type III, IV).
9. Absence of fixed or removable orthodontic appliance or removable partial dentures;
10. Able to read and understand the local language;
11. Male or non-pregnant, non-lactating female, by self-report;
12. Male and female subjects with reproductive potential must agree to practice a medically acceptable form of birth control during the study and for 30 days following the last dose of investigational product. Females must have used such birth control for at least 3 months prior to the Baseline visit.

    Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include:
    * Abstinence from reproductive intercourse when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;
    * Established use of hormonal methods of contraception (oral, injected, implanted, patch or vaginal ring);
    * Intrauterine device (IUD) or intrauterine system (IUS);
    * Barrier methods of contraception with spermicide: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository;
    * Surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy); and
    * A female subject who is postmenopausal (i.e., amenorrheic for at least 12 months prior to the Baseline visit) is not considered of reproductive potential.
13. Willing for this to be the only investigational product used during this time period; and
14. Willing and able to comply with all study procedures and attend the scheduled visits for the duration of the study.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes and mouth rinses and red food dye;
2. Dental prophylaxis within 2 weeks prior to Screening visit;
3. Antibiotic, anti-inflammatory or anticoagulant therapy during the study or within one month prior to the baseline exam;
4. Regular use of chemotherapeutic antiplaque/antigingivitis products such as triclosan, essential oil, cetylpyridinium chloride, or chlorhexidine containing mouth rinses within three weeks prior to baseline;
5. Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results);
6. Significant unstable or uncontrolled medical condition which may interfere with a subject's participation in the study, at the discretion of the Investigator;
7. Participation in any other clinical study within 30 days of Visit 1;
8. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each); and
9. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, substance or alcohol abuse or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maher Naji, D.D.S, Principal Investigator — All Sum Research Center Ltd.
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Control (W002194-221P): Negative Control - 5% Hydroalcohol Mouth Rinse (20 mL) twice daily after brushing
- 19292-116A: Cool Mint® Listerine® Antiseptic Mouth Rinse (20 mL) twice daily after brushing
- 11965-059: Listerine® Zero™ Mouth Rinse (20 mL) twice daily after brushing
Period: Overall Study
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Started | 53 | 52 | 53
Completed | 53 | 52 | 53
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059 | Total
Number analyzed (Participants) | 53 | 52 | 53 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.97) | 41.7 (12.48) | 45.5 (11.18) | 44.5 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 32 | 100
  Male | 14 | 23 | 21 | 58
Region of Enrollment [Number; unit: participants]
  Canada | 53 | 52 | 53 | 158

OUTCOME MEASURES:

1. Primary Outcome: Whole Mouth Mean Modified Gingival Index (MGI) at Week 3
Description: Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth according to the following scale: 0: Normal (absence of inflammation), 1: Mild inflammation (slight change in color, little change in texture) of any portion of the gingival unit, 2: Mild inflammation of the entire gingival unit, 3: Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit, and 4: Severe inflammation marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. The score for each participant was calculated by averaging their tooth site scores at Week 3.
Time Frame: 3 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized participants who used at least one dose of the study product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
units on a scale | 2.004 (0.0114) | 1.770 (0.0115) | 1.807 (0.0113)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — Per statistical analysis plan, Hochberg's method at significance level 0.05 was applied to jointly evaluate Whole Mouth Mean MGI at Wk 3 and Whole Mouth Mean PI at Wk 3 for both Listerine rinses vs control. Family-wise error controlled at 0.05; Terms included treatment with baseline whole mouth mean modified gingival index as a covariate; Least Squares Mean Difference = -0.234, 95% CI 2-sided [-0.266 to -0.202], Standard Error of Mean 0.0162
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Terms included treatment with baseline whole mouth mean modified gingival index as a covariate; Least Squares Mean Difference = -0.197, 95% CI 2-sided [-0.228 to -0.165], Standard Error of Mean 0.0161

2. Primary Outcome: Whole Mouth Mean Plaque Index (PI) at Week 3
Description: Plaque area was measured based on the Turesky modification of the Quigley-Hein Plaque Index and was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) of all scorable teeth, following disclosing, according to the following scale: 0: No plaque, 1: Separate flecks or discontinuous band of plaque at the gingival (cervical) margin, 2: Thin (up to 1 mm), continuous band of plaque at the gingival margin, 3: Band of plaque wider than 1 mm but less than 1/3 of surface, 4: Plaque covering 1/3 or more, but less than 2/3 of surface, 5: Plaque covering 2/3 or more of surface. The score for each participant was calculated by averaging their tooth site scores at Week 3.
Time Frame: 3 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
units on a scale | 2.434 (0.0202) | 1.965 (0.0204) | 2.055 (0.0202)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Terms included treatment with baseline whole mouth mean plaque index as a covariate; Least Squares Mean Difference = -0.469, 95% CI 2-sided [-0.526 to -0.413], Standard Error of Mean 0.0286
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Terms included treatment with baseline whole mouth mean plaque index as a covariate; Least Squares Mean Difference = -0.379, 95% CI 2-sided [-0.435 to -0.322], Standard Error of Mean 0.0286

3. Secondary Outcome: Whole Mouth Mean Gingival Bleeding Index (BI) at Week 3
Description: Bleeding was assessed using a periodontal probe with a 0.5 mm diameter tip which was inserted into the gingival crevice, and swept from distal to mesial, around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 4 gingival areas (disto-buccal, midbuccal, mid-lingual, and mesio-lingual) around each tooth was assessed. After approximately 30 seconds, bleeding at each gingival unit was recorded according to the following scale: 0: Absence of bleeding after 30 seconds, 1: Bleeding after 30 seconds, and 2: Immediate bleeding. The score for each participant was calculated by averaging their tooth site scores at Week 3.
Time Frame: 3 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
units on a scale | 0.098 (0.0042) | 0.067 (0.0042) | 0.072 (0.0042)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment with baseline whole mouth mean gingival bleeding index as a covariate; Least Squares Mean Difference = -0.030, 95% CI 2-sided [-0.042 to -0.019], Standard Error of Mean 0.0060
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment with baseline whole mouth mean gingival bleeding index as a covariate; Least Squares Mean Difference = -0.026, 95% CI 2-sided [-0.038 to -0.014], Standard Error of Mean 0.0059

4. Secondary Outcome: Change From Baseline in the Percentage of Healthy Sites (Modified Gingival Index (MGI) Scores of 0 or 1) at Week 3
Description: Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth according to the following scale: 0: Normal (absence of inflammation), 1: Mild inflammation (slight change in color, little change in texture) of any portion of the gingival unit, 2: Mild inflammation of the entire gingival unit, 3: Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit, and 4: Severe inflammation marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. The score for each participant was the change from baseline in the percentage of sites with an MGI score of 0 or 1 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of MGI scores of 0 or 1
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of MGI scores of 0 or 1 | 5.5 (4.52) | 27.5 (9.45) | 24.3 (8.68)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; The null hypothesis was no difference between treatment groups. The alternative hypothesis was a difference between treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 23.240, 95% CI 2-sided [20.75 to 25.85] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 19.444, 95% CI 2-sided [17.09 to 22.22] — 95% Confidence limits for the location shift

5. Secondary Outcome: Change From Baseline in the Percentage of Virtually Plaque-Free Sites (Plaque Index (PI) Scores of 0 or 1) at Week 3
Description: Plaque area was measured based on the Turesky modification of the Quigley-Hein Plaque Index and was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) of all scorable teeth, following disclosing, according to the following scale: 0: No plaque, 1: Separate flecks or discontinuous band of plaque at the gingival (cervical) margin, 2: Thin (up to 1 mm), continuous band of plaque at the gingival margin, 3: Band of plaque wider than 1 mm but less than 1/3 of surface, 4: Plaque covering 1/3 or more, but less than 2/3 of surface, 5: Plaque covering 2/3 or more of surface. The score for each participant was the change from baseline in the percentage of sites with a PI score of 0 or 1 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PI scores of 0 or 1
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of PI scores of 0 or 1 | 3.2 (3.60) | 20.9 (10.76) | 18.3 (9.55)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 19.048, 95% CI 2-sided [15.94 to 21.73] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 15.939, 95% CI 2-sided [12.50 to 18.67] — 95% Confidence limits for the location shift

6. Secondary Outcome: Change From Baseline in the Percentage of Non-Bleeding Sites (Gingival Bleeding Index (BI) Scores of 0) at Week 3
Description: Bleeding was assessed using a periodontal probe with a 0.5 mm diameter tip which was inserted into the gingival crevice, and swept from distal to mesial, around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 4 gingival areas (disto-buccal, midbuccal, mid-lingual, and mesio-lingual) around each tooth was assessed. After approximately 30 seconds, bleeding at each gingival unit was recorded according to the following scale: 0: Absence of bleeding after 30 seconds, 1: Bleeding after 30 seconds, and 2: Immediate bleeding. The score for each participant was the change from baseline in the percentage of sites with a BI score of 0 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of BI scores of 0
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of BI scores of 0 | 0.3 (2.30) | 2.5 (2.66) | 2.1 (3.17)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 2.050, 95% CI 2-sided [1.30 to 2.78] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 1.190, 95% CI 2-sided [0.93 to 2.06] — 95% Confidence limits for the location shift

7. Secondary Outcome: Change From Baseline in the Percentage of Problem Sites (Modified Gingival Index (MGI) Scores of ≥ 3) at Week 3
Description: Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth according to the following scale: 0: Normal (absence of inflammation), 1: Mild inflammation (slight change in color, little change in texture) of any portion of the gingival unit, 2: Mild inflammation of the entire gingival unit, 3: Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit, and 4: Severe inflammation marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. The score for each participant was the change from baseline (i.e., Baseline Score minus Week 3 Score) in the percentage of sites with an MGI score ≥3 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of MGI scores of >= 3
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of MGI scores of >= 3 | -0.6 (4.34) | 0.9 (4.15) | 0.3 (3.85)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.016, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 1.316, 95% CI 2-sided [0.00 to 2.78] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.197, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 0.926, 95% CI 2-sided [-0.16 to 1.85] — 95% Confidence limits for the location shift

8. Secondary Outcome: Change From Baseline in the Percentage of Problem Sites (Plaque Index (PI) Scores of ≥ 3) at Week 3
Description: Plaque area was measured based on the Turesky modification of the Quigley-Hein Plaque Index and was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) of all scorable teeth, following disclosing, according to the following scale: 0: No plaque, 1: Separate flecks or discontinuous band of plaque at the gingival (cervical) margin, 2: Thin (up to 1 mm), continuous band of plaque at the gingival margin, 3: Band of plaque wider than 1 mm but less than 1/3 of surface, 4: Plaque covering 1/3 or more, but less than 2/3 of surface, 5: Plaque covering 2/3 or more of surface. The score for each participant was the change from baseline (i.e., Baseline Score minus Week 3 Score) in the percentage of sites with a PI score ≥3 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PI scores of >= 3
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of PI scores of >= 3 | 0.1 (13.12) | 23.5 (14.45) | 18.9 (13.84)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 23.214, 95% CI 2-sided [18.21 to 28.77] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 18.590, 95% CI 2-sided [13.69 to 23.81] — 95% Confidence limits for the location shift

9. Secondary Outcome: Change From Baseline in the Percentage of Problem Sites (Plaque Index (PI) Scores of ≥ 2) at Week 3
Description: Plaque area was measured based on the Turesky modification of the Quigley-Hein Plaque Index and was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) of all scorable teeth, following disclosing, according to the following scale: 0: No plaque, 1: Separate flecks or discontinuous band of plaque at the gingival (cervical) margin, 2: Thin (up to 1 mm), continuous band of plaque at the gingival margin, 3: Band of plaque wider than 1 mm but less than 1/3 of surface, 4: Plaque covering 1/3 or more, but less than 2/3 of surface, 5: Plaque covering 2/3 or more of surface. The score for each participant was the change from baseline (i.e., Baseline Score minus Week 3 Score) in the percentage of sites with a PI score ≥2 at Week 3.
Time Frame: Baseline to 3 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PI scores of >= 2
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Number analyzed (Participants) | 53 | 52 | 53
percentage of PI scores of >= 2 | 3.2 (3.60) | 20.9 (10.76) | 18.3 (9.55)
Statistical Analysis 1: Comparison: Negative Control (W002194-221P) vs 19292-116A; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 19.048, 95% CI 2-sided [15.94 to 21.73] — 95% Confidence limits for the location shift
Statistical Analysis 2: Comparison: Negative Control (W002194-221P) vs 11965-059; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; P-values were based on Wilcoxon Rank Sum Test on the change from baseline; Hodges-Lehmann estimate of difference = 15.939, 95% CI 2-sided [12.50 to 18.67] — 95% Confidence limits for the location shift

ADVERSE EVENTS:
Time Frame: Day 22 ± 2 days, + 30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 3 (Day 22 ± 2 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Negative Control (W002194-221P) | 19292-116A | 11965-059
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.